CLINICAL TRIAL: NCT04711356
Title: An Open Label Study to Evaluate the Safety and Immunogenicity of an Ad26.ZEBOV Booster Dose in Children Previously Vaccinated With the Ad26.ZEBOV and MVA-BN-Filo Vaccine Regimen
Brief Title: Ad26.ZEBOV Booster in Children Previously Vaccinated With Ad26.ZEBOV and MVA-BN-Filo (EBOVAC Booster Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Innovative Medicines Initiative (Other); University of Sierra Leone (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAC52150EBL2011
Record Dates: First submitted 2020-12-09; First posted 2021-01-15 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2021-10

CONDITIONS: Ebola Virus Disease
Keywords: Ad26.ZEBOV; booster vaccination; children
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Intervention Model Description: All participants will receive a single dose of Ad26.ZEBOV at a dose of 5x10^10 viral particles (vp) administered intramuscularly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Intervention (Experimental): All study participants will receive an Ad26.ZEBOV vaccine at a dose of 5x10^10 vp given via IM injection
  Interventions: Drug: Ad26.ZEBOV booster vaccination, given at a dose of 5x10^10 vp, via IM injection

INTERVENTIONS:
Drug: Ad26.ZEBOV booster vaccination, given at a dose of 5x10^10 vp, via IM injection — Ad26.ZEBOV is a monovalent, replication-incompetent adenovirus serotype 26-based vector that expresses the full-length Ebola virus Mayinga glycoprotein

SUMMARY:
This is an open-label study evaluating the safety and immunogenicity of a booster dose of Ad26.ZEBOV administered to children who were previously vaccinated with Ad26.ZEBOV followed by MVA-BN-Filo 56 days later.

DETAILED DESCRIPTION:
RATIONALE:

Over 600 children have received the adenovirus serotype 26 expressing the Ebola virus Mayinga glycoprotein (Ad26.ZEBOV), modified Vaccinia Ankara Bavarian Nordic vector expressing multiple filovirus proteins (MVA- BN-Filo) Ebola vaccine regimen in the EBL2002 and EBL3001 clinical trials. The vaccine regimen was well tolerated and highly immunogenic in children; however, the durability of vaccine-induced immune responses is not known. In adults previously vaccinated with the Ad26.ZEBOV and MVA-BN-Filo regimen, a booster vaccination with Ad26.ZEBOV was safe and induced a strong anamnestic response within seven days of the booster vaccination. It is important to establish if a booster dose of Ad26.ZEBOV is safe and immunogenic also in children, as this can guide the clinical use of the Ad26.ZEBOV, MVA-BN-Filo vaccine regimen in this age group. For example, it could support the strategy of boosting immunised children at the start of an Ebola outbreak.

STUDY OBJECTIVES AND HYPOTHESIS:

This study aims to evaluate the safety and immunogenicity of an Ad26.ZEBOV booster dose in healthy children who were previously (>2 years) vaccinated with the Ad26.ZEBOV (dose 1) followed by MVA-BN-Filo (dose 2) 56 days later, by monitoring adverse events (AEs) following the booster vaccination and by assessing binding antibody responses using the Filovirus Animal Non-Clinical Group (FANG) Enzyme-Linked Immunosorbent Assay (ELISA).

Primary Objectives:

* To assess the safety and tolerability of a booster dose of Ad26.ZEBOV at a dose of 5x10^10 viral particles (vp) in children previously vaccinated with the Ad26.ZEBOV, MVA-BN-Filo vaccine regimen with a 56-day interval. Safety and tolerability will be assessed by measuring:

  1. Incidence of solicited local (at the administration site) and systemic adverse events as assessed on the day of booster vaccination and by diary card for 7 days after booster vaccination.
  2. Incidence of unsolicited adverse events from the day of the booster vaccination to 28 days post booster vaccination.
* To assess vaccine-induced humoral immune responses to the Ebola virus glycoprotein (EBOV GP), as measured by FANG ELISA (EU/ml), at 7 and 21 days following a booster dose of Ad26.ZEBOV at a dose of 5x10^10 vp in children previously vaccinated with the Ad26.ZEBOV, MVA-BN-Filo vaccine regimen with a 56-day interval.

Exploratory Objectives

• To assess neutralising antibody responses directed against the Ad26 vector before booster vaccination as measured by a virus neutralization assay (VNA).

Hypothesis: as this study is designed to provide descriptive information regarding safety and immunogenicity without formal treatment comparisons, no formal statistical hypothesis testing is planned.

OVERVIEW OF THE STUDY:

This is an open-label study evaluating the immune response to a booster dose of Ad26.ZEBOV administered to children who were previously vaccinated with Ad26.ZEBOV followed by MVA-BN-Filo 56 days later. Only subjects who received the Ad26.ZEBOV and MVA-BN-Filo regimen during their participation in the VAC52150EBL3001 (EBOVAC-Salone) vaccine trial (ClinicalTrials.gov Identifier: NCT02509494), are eligible for enrolment in this study. Participants will be recruited in two age groups: children aged 4-11 years at the time of dose 1 vaccination and children aged 1-3 years at the time of dose 1 vaccination in the EBOVAC-Salone trial. Approximately 25 subjects will be enrolled in each of these two age groups. Parents/guardians will be asked to consent for the participation of their children in the study. Children aged 7 years and older at the time of enrolment in this study will be asked to give positive assent for their participation. Participants will be followed up to 28 days after their booster vaccination. The study will be conducted in Kambia, Sierra Leone.

Study Population: potential participants must be healthy children (based on physical examination, medical history, a haematological assessment and clinical judgment) who received the Ad26.ZEBOV and MVA-BN-Filo vaccine regimen in the EBOVAC-Salone trial and were aged ≥1 to ≤11 years at the time of dose 1 vaccination. They must also be enrolled in the long-term follow-up study to the EBOVAC-Salone trial, VAC52150EBL3005 (EBOVAC-Salone Extension study, ClinicalTrials.gov Identifier: NCT03820739) but not in the immunogenicity subset.

Dosage and administration: a single dose of Ad26.ZEBOV at a dose of 5x10^10 vp administered intramuscularly.

Safety evaluations: solicited local (at the administration site) and systemic AEs will be assessed on the day of vaccination and using a diary for a period of 7 days following the booster vaccination. Unsolicited AEs will be tracked for 28 days following booster vaccination, while serious adverse events will be tracked for the duration of the study.

Immunogenicity evaluations: blood will be drawn for assessments of immune responses at 7 and 21 days post booster vaccination.

STATISTICAL METHODS:

The primary analysis will be done when all subjects have completed their 28-day post-booster visit or discontinued earlier. This analysis will include all available data up to this point.

Sample Size Determination: the sample size is a convenience sample and is not based on formal hypothesis testing considerations.

Safety analysis: no formal statistical testing of safety data is planned. Safety data will be analysed descriptively by age group, 1-3 years and 4-11 years (age the participant was when they received dose 1 vaccination in the EBOVAC-Salone trial).

Immunogenicity analysis: no formal hypothesis on immunogenicity will be tested. Descriptive statistics (i.e. geometric mean and 95% confidence interval, as appropriate) will be calculated for continuous immunologic parameters at all available time points. Graphical representations of immunologic parameters will be made as applicable.

Frequency tabulations will be calculated for discrete (qualitative) immunologic parameters (i.e. responder rate), as applicable. Responders rate defined as >2.5-time increase over baseline value (or lower limit of quantitation [LLOQ]) pre-dose 1 vaccination in the EBOVAC-Salone trial, will be calculated depending on availability of sample results from the EBOVAC-Salone trial.

ELIGIBILITY:
Inclusion Criteria:

1. Child must be enrolled in the VAC52150EBL3005 (EBOVAC-Salone Extension) study but not in the immunogenicity subset of EBOVAC-Salone Extension study.
2. Child must be a former participant in the VAC52150EBL3001 (EBOVAC-Salone) trial, and have received Ad26.ZEBOV (dose 1) vaccination followed by the MVA-BN-Filo (dose 2) vaccination within the EBOVAC- Salone trial window for dose 2 vaccination.
3. Child must have been aged 1 to 11 years old at the time of dose 1 vaccination in the EBOVAC-Salone trial.
4. The parent/guardian must consent for their child to participate in the VAC52150EBL2011 study. Children aged 7 years and older will be asked to give positive assent for their participation in the study.
5. The parent/guardian is willing/able to ensure that their child adheres to the prohibitions and restrictions specified in this protocol.
6. Child must be healthy in the investigator's clinical judgement (and the parent/guardian's judgement) on the basis of medical history, physical examination, vital signs, and a haematological assessment (i.e. full blood count) performed at screening. Subjects must meet the following haematology parameters within 28 days before Day 1:

   * Haemoglobin ≥8.0 g/dL for children aged 1 to <5 years, ≥9g/dL for children aged 5 or older
   * Platelet count ≥100 x 10^9/L
   * White blood cell count ≥5.0 x 10^9/L
7. Adolescent girls who have started their menstrual periods and/or are ≥12 years of age at the time of screening, must have a negative urine β-hCG pregnancy test at screening and immediately prior to the booster vaccination on Day 1.
8. The parent/guardian is available and willing to have their infant participate for the duration of the study visits.
9. The parent/guardian must have a means to be contacted.
10. The parent/guardian must pass the Test of Understanding (TOU)

Exclusion Criteria:

1. Participants in the EBOVAC-Salone trial who were allocated to the control arm receiving the WHO- prequalified Meningococcal Group A, C, W135 and Y conjugate vaccine.
2. Participants in the EBOVAC-Salone trial who were age 12 years and older at the time of dose 1 vaccination.
3. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccine, e.g., polysorbate 80, ethylenediaminetetraacetic acid or L-histidine for Ad26.ZEBOV vaccine), including known allergy to chicken or egg proteins and aminoglycosides (gentamicin).
4. Presence of acute illness (this does not include minor illnesses such as mild diarrhoea or mild upper respiratory tract infection) or axillary temperature ≥38C on Day 1. Participants with such symptoms will be excluded from enrolment at that time but may be rescheduled for enrolment at a later date within the screening window.
5. Clinically significant history of skin disorder (e.g., psoriasis, contact dermatitis), allergy, symptomatic immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness as judged by the investigator or other delegated individual.
6. Adolescent girls who are known to be pregnant or breastfeeding at screening.
7. Received a blood transfusion or other blood products within 8 weeks of vaccination day.
8. Children who have been vaccinated with live-attenuated vaccines within 30 days before the study vaccination, and with inactivated vaccine within 15 days before the study vaccination.
9. Children who, in the opinion of the investigator, are unlikely to adhere to the requirements of the study or are unlikely to complete the vaccination and observation.
10. Any other finding which in the opinion of the investigator or other delegated individual would increase the risk of an adverse outcome from participation in the study.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Watson-Jones, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Bailah Leigh, MD, Principal Investigator — University of Sierra Leone
Locations (1):
- EBOVAC Kambia 1 clinic, Kambia, Sierra Leone

IPD SHARING:
Plan to Share IPD: Yes
The clinical trial results will be published in an open access, peer-reviewed journal, which will include the study protocol. A summary of the study results will be included within the trial registration record in PACTR and ClinicalTrials.gov
  Following publication of the primary and exploratory objectives as detailed in the protocol, individual de-identified participants' data and a data dictionary will be made available upon request via the London School of Hygiene & Tropical Medicine research data repository, LSHTM Data Compass at http://datacompass.lshtm.ac.uk. Requests with a defined analysis plan can be sent via LSHTM Data Compass.
Supporting Information: Study Protocol
Time Frame: within 12 months of the study completion date
Access Criteria: open

REFERENCES:
- [Derived] Manno D, Bangura A, Baiden F, Kamara AB, Ayieko P, Kallon J, Foster J, Conteh M, Connor NE, Koroma B, Njie Y, Borboh P, Keshinro B, Lawal BJ, Kroma MT, Otieno GT, Deen AT, Choi EM, Balami AD, Gaddah A, McLean C, Luhn K, Adetola HH, Deen GF, Samai M, Lowe B, Robinson C, Leigh B, Greenwood B, Watson-Jones D. Safety and immunogenicity of an Ad26.ZEBOV booster dose in children previously vaccinated with the two-dose heterologous Ad26.ZEBOV and MVA-BN-Filo Ebola vaccine regimen: an open-label, non-randomised, phase 2 trial. Lancet Infect Dis. 2023 Mar;23(3):352-360. doi: 10.1016/S1473-3099(22)00594-1. Epub 2022 Oct 20. PMID 36273490

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened between 8 July and 18 August 2021 at one clinic in Kambia Town, located in Kambia District in the North West Province of Sierra Leone.
Pre-assignment Details: All the enrolled participants received the study intervention.
Groups:
- Study Intervention: Ad26.ZEBOV booster vaccination at a dose of 5x10^10 vp, via IM injection
Period: Overall Study
Arm/Group | Study Intervention
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Intervention
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6 [4 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Sierra Leone | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local (at the Administration Site) Adverse Events
Description: Number and percentage of participants with at least one solicited local adverse event (i.e. pain, erythema, pruritus and swelling)
Time Frame: From the booster vaccination to 7 days post booster
Population: All participants who had received the Ad26.ZEBOV booster
Measure: Count of Participants; unit: Participants
Arm/Group | Study Intervention
Number analyzed (Participants) | 50
Participants | 18

2. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events
Description: Number and percentage of participants with at least one solicited systemic adverse event (i.e. arthralgia, chills, fatigue, headache, myalgia, nausea and pyrexia)
Time Frame: From the booster vaccination to 7 days post booster
Population: All participants who had received the Ad26.ZEBOV booster
Measure: Count of Participants; unit: Participants
Arm/Group | Study Intervention
Number analyzed (Participants) | 50
Participants | 16

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Number and percentage of participants with at least one unsolicited adverse event
Time Frame: From the booster vaccination to 28 days post booster
Population: All participants who had received the Ad26.ZEBOV booster
Measure: Count of Participants; unit: Participants
Arm/Group | Study Intervention
Number analyzed (Participants) | 50
Participants | 32

4. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Number and percentage of participants with serious adverse events
Time Frame: From the booster vaccination to 28 days post booster
Population: All participants who had received the Ad26.ZEBOV booster
Measure: Count of Participants; unit: Participants
Arm/Group | Study Intervention
Number analyzed (Participants) | 50
Participants | 0

5. Primary Outcome: Pre-booster Baseline Humoral Immune Responses to the Ebola Virus Glycoprotein (EBOV GP)
Description: EBOV GP antibody geometric mean concentration measured by FANG ELISA in Elisa Units (EU) per millilitre
Time Frame: day 1 before booster administration
Population: All boosted participants who had at least one evaluable post-booster sample and had no major protocol deviations that could have influenced the immune response after booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Study Intervention
Number analyzed (Participants) | 49
ELISA units/mL | 640 [461 to 888]

6. Primary Outcome: Vaccine-induced Humoral Immune Responses to the Ebola Virus Glycoprotein (EBOV GP)
Description: EBOV GP antibody geometric mean concentration measured by FANG ELISA in Elisa Units (EU) per millilitre
Time Frame: At 7 days post booster
Population: All boosted participants who had an evaluable post-booster sample and had no major protocol deviations that could have influenced the immune response after booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Study Intervention
Number analyzed (Participants) | 50
ELISA units/mL | 28561 [20255 to 40272]

7. Primary Outcome: Vaccine-induced Humoral Immune Responses to the Ebola Virus Glycoprotein (EBOV GP)
Description: EBOV GP antibody geometric mean concentration measured by FANG ELISA in Elisa Units (EU) per millilitre
Time Frame: At 21 days post booster
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Study Intervention
Number analyzed (Participants) | 49
ELISA units/mL | 64690 [48356 to 86541]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events were recorded from the booster vaccination (day 1) to 7 days after the booster vaccination (day 8) Unsolicited adverse events were recorded from the booster vaccination (day 1) to 28 days after the booster vaccination (day 29)
Description: Participants were observed for at least 30 minutes after vaccination. During the first 7 days post booster, field workers visited participants at home daily to record local and systemic solicited AEs using a diary card. Parents or guardians of participants received a 24-hour phone number to contact in case of medical problems and were asked about the participant's health at every study visit. Unsolicited AEs were recorded from the booster vaccination until 28 days post-booster vaccination.
Arm/Group | Study Intervention
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 32/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Intervention (N=50)
Malaria (Infections and infestations) | 25 (25) — Unsolicited adverse event
Upper respiratory tract infections (Infections and infestations) | 7 (7) — Unsolicited adverse event
Lower respiratory tract infection/pneumonia (Infections and infestations) | 4 (4) — Unsolicited adverse event
Rhinitis (Infections and infestations) | 1 (1) — Unsolicited adverse event
Worm infestation (Infections and infestations) | 2 (2) — Unsolicited adverse event
Acute otitis media (Infections and infestations) | 1 (1) — Unsolicited adverse event
Scabies (Infections and infestations) | 2 (2) — Unsolicited adverse event
Urinary tract infection (Infections and infestations) | 2 (2) — Unsolicited adverse event
Gastroenteritis (Infections and infestations) | 1 (1) — Unsolicited adverse event
Thrombocytopaenia (Blood and lymphatic system disorders) | 1 (1) — Unsolicited adverse event
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) — Unsolicited adverse event
Leg ulcer (Vascular disorders) | 1 (1) — Unsolicited adverse event
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Unsolicited adverse event
Eye burns (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited adverse event
Dental caries (Gastrointestinal disorders) | 1 (1) — Unsolicited adverse event
Swollen thumb (General disorders) | 1 (1) — Unsolicited adverse event
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) — Solicited local adverse events (at the injection site)
Pain (Skin and subcutaneous tissue disorders) | 18 (18) — Solicited local adverse events (at the injection site)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Solicited local adverse events (at the injection site)
Swelling (Skin and subcutaneous tissue disorders) | 0 (0) — Solicited local adverse events (at the injection site)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) — Solicited systemic adverse events
Chills (General disorders) | 6 (6) — Solicited systemic adverse events
Fatigue (General disorders) | 8 (8) — Solicited systemic adverse events
Headache (General disorders) | 11 (11) — Solicited systemic adverse events
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) — Solicited systemic adverse events
Nausea (Gastrointestinal disorders) | 3 (3) — Solicited systemic adverse events
Pyrexia (General disorders) | 6 (6) — Solicited systemic adverse events

LIMITATIONS AND CAVEATS:
In the study protocol, the follow-up was only 28 days due to the end of the grant that funded the study.

Neutralising antibodies and cellular immune responses post booster could not be assessed within the timeframe of the grant and were not included in the protocol.

We do not know if the concentrations of binding antibodies achieved after booster vaccination indicate protection against Ebola virus disease because an antibody threshold correlating with protection has not yet been established.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT04711356/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT04711356/SAP_001.pdf